CLINICAL TRIAL: NCT06179004
Title: Randomized Controlled Trial of Supraclavicular Bupivacaine Vs. Supraclavicular Liposomal Bupivacaine for Orthopedic Wrist Surgery
Brief Title: Supraclavicular Bupivacaine Vs. Supraclavicular Liposomal Bupivacaine for Orthopedic Wrist Surgery
Acronym: Vs
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-1116
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Distal Radius Fractures; Wrist Fractures
MeSH Terms: conditions — Wrist Fractures | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Interim analysis will be performed when data collection is complete for 40 participants.
Who Masked: Participant, Investigator
Masking Description: As participants are enrolled in this study, a study identification will be created as their basic demographic information is entered into the secure RedCap database. At this time, the RedCap randomization tool will randomize the subject to either group 1 or 2.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Supraclavicular Liposomal Bupivacaine group (Experimental): This group will receive the liposomal bupivacaine
  Interventions: Drug: Liposomal bupivacaine
- Supraclavicular Plain Bupivacaine group (Active Comparator): This group will receive the plain bupivacaine
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Liposomal bupivacaine — 133mg Liposomal bupivacaine plus 10mL 0.5% bupivacaine administered in a supraclavicular single shot perineural injection
  Other Names: Exparel
  Arms: Supraclavicular Liposomal Bupivacaine group
Drug: Bupivacaine Hydrochloride — 20mL 0.25% bupivacaine administered in a supraclavicular single shot perineural injection
  Arms: Supraclavicular Plain Bupivacaine group

SUMMARY:
Orthopedic wrist procedures often cause significant postoperative pain. A supraclavicular nerve block is an effective and proven method to help reduce postoperative pain and decrease opioid use around the time of upper extremity surgery. Liposomal bupivacaine (Exparel) has been approved for use around the brachial plexus, but its analgesic efficacy has limited data. The investigators' goal is to evaluate the effectiveness of Exparel as compared to plain bupivacaine. The investigators hope to ensure the quality of pain control around the time of distal radius fracture repair and reduce the variability of care at the investigators institution by prospectively and rigorously collecting perioperative data during this study.

DETAILED DESCRIPTION:
Purpose: Orthopedic wrist procedures often cause significant postoperative pain. A supraclavicular nerve block is an effective and proven method to help reduce postoperative pain and decrease opioid use around the time of shoulder surgery. Liposomal bupivacaine (Exparel) has been approved for use around the brachial plexus, but its analgesic efficacy has limited data. The investigators goal is to evaluate the effectiveness of Exparel as compared to the investigators prior standard practice of using plain bupivacaine. The investigators hope to ensure the quality of pain control around the time of distal radius fracture repair and reduce the variability of care at the investigators institution by prospectively and rigorously collecting perioperative data during this study.

Participants: Adult participants age > 18 undergoing orthopedic wrist surgery at the University of North Carolina ambulatory surgery center and University of North Carolina Hillsborough campus Exclusion Criteria: the below are simply contraindications to regional anesthesia in general, this is a pragmatic study to evaluate the quality of care for these subjects with no additional exclusion criteria.- Contraindications to regional anesthesia- Significant peripheral neuropathy or neurological disorder affecting the upper extremity- Pregnancy- Cognitive or psychiatric condition that might affect patient assessment and/or inability to provide informed consent.

Procedures (methods): This is a prospective, randomized comparison of participants undergoing orthopedic wrist procedures that receive one of two types of supraclavicular nerve block. Group 1 will be comprised of patients with a preoperative supraclavicular nerve block placed with 20 mL 0.5% bupivacaine. Group 2 will be comprised of participants with a preoperative supraclavicular nerve block placed with 10 mL 0.5% bupivacaine and 10 mL 1.3% Liposomal Bupivacaine (Exparel). All subjects in both groups will have a similar intraoperative general anesthetic with multimodal analgesic pre-op oral medications. Outcomes measured by Post anesthesia care unit assessment and telephone follow up: see uploaded data collection form.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* Scheduled for orthopedic wrist surgery at University of North Carolina at Chapel Hill.

Exclusion Criteria:

* Contraindications to regional anesthesia
* Emergent surgery Open fractures will be treated emergently and will not allow adequate lead time for enrollment in this study. Also, open fractures are usually accompanied by other traumatic injuries that would confound the pain related outcomes in this study.
* Significant peripheral neuropathy or neurological disorder affecting the upper extremity
* Pregnancy Pregnant women have physiologic changes that make them more sensitive to local anesthetics. That would introduce a confounding element in interpreting the effectiveness of the peripheral nerve blocks being studied.
* Cognitive or psychiatric condition that might affect patient assessment and/or inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pre-operative and 48-hour Post-operative Quality of Recovery 15 survey score | Pre-operative and at 24 hours and 48 hours post-operative
  The quality of recovery-15 (QoR-15) is a validated questionnaire to assess postoperative recovery. Scale is based on 15 questions, each question score range is 0-10 (0 being poor and 10 being excellent) The survey will be conducted at 24 hours intervals after surgery up to 48 hours total after surgery. The total score range is 0-150, where a score of 0 would be the worst possible score, and 150 would be the best possible score

SECONDARY OUTCOMES:
Difference in Participant Reported Pain Scores | Post-operative period up to 48 hours after surgery
  These pain scores will be collected immediately after surgery in the recovery room, and on postoperative days 1 and 2 during follow up telephone encounters. The estimate of interest is the difference in patient reported pain scores (numeric 0-10) between groups at these points in time.
Time to First Dose of Opioid Medication | Post-operative period up to 48 hours after surgery
  Investigate opioid medication consumption by recording time to first opioid medication administered.
Total opioid dose through Post-op Day 2 | Post-operative period up to 48 hours after surgery
  Investigate opioid medication consumption by recording total opioid dose for each group through postoperative day 2.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Schoenherr, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abell DJ, Barrington MJ. Pneumothorax after ultrasound-guided supraclavicular block: presenting features, risk, and related training. Reg Anesth Pain Med. 2014 Mar-Apr;39(2):164-7. doi: 10.1097/AAP.0000000000000045. PMID 24496168
- [Result] Brown CA, Ghanouni A, Williams R, Payne SH, Ghareeb PA. Safety and Efficacy of Liposomal Bupivacaine Supraclavicular Nerve Blocks in Open Treatment of Distal Radius Fractures: A Perioperative Pain Management Protocol. Ann Plast Surg. 2023 Jun 1;90(6S Suppl 4):S332-S336. doi: 10.1097/SAP.0000000000003464. Epub 2023 Jan 31. PMID 36752544
- [Result] Hussain N, Brull R, Sheehy B, Essandoh MK, Stahl DL, Weaver TE, Abdallah FW. Perineural Liposomal Bupivacaine Is Not Superior to Nonliposomal Bupivacaine for Peripheral Nerve Block Analgesia. Anesthesiology. 2021 Feb 1;134(2):147-164. doi: 10.1097/ALN.0000000000003651. PMID 33372953
- [Result] Myles PS, Shulman MA, Reilly J, Kasza J, Romero L. Measurement of quality of recovery after surgery using the 15-item quality of recovery scale: a systematic review and meta-analysis. Br J Anaesth. 2022 Jun;128(6):1029-1039. doi: 10.1016/j.bja.2022.03.009. Epub 2022 Apr 14. PMID 35430086
- [Result] Rundgren J, Mellstrand Navarro C, Ponzer S, Regberg A, Serenius S, Enocson A. Regional or General Anesthesia in the Surgical Treatment of Distal Radial Fractures: A Randomized Clinical Trial. J Bone Joint Surg Am. 2019 Jul 3;101(13):1168-1176. doi: 10.2106/JBJS.18.00984. PMID 31274718
- [Result] Schoenherr JW, Gonzalez M, Serrano R, Park M, Lee Z, Cobb K, Howard C, Flynn D, Li Q, Grant S, Bullard T. Quality of Recovery After Rotator Cuff Repair With Interscalene Liposomal Bupivacaine Versus Interscalene Nerve Catheter. Orthop J Sports Med. 2022 Nov 22;10(11):23259671221134819. doi: 10.1177/23259671221134819. eCollection 2022 Nov. PMID 36458106
- [Result] Chazapis M, Walker EM, Rooms MA, Kamming D, Moonesinghe SR. Measuring quality of recovery-15 after day case surgery. Br J Anaesth. 2016 Feb;116(2):241-8. doi: 10.1093/bja/aev413. PMID 26787793
- [Result] D'Souza RS, Johnson RL. Supraclavicular Block. [Updated 2023 Jan 8]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2023 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK519056/
- [Result] Myles PS, Myles DB, Galagher W, Chew C, MacDonald N, Dennis A. Minimal Clinically Important Difference for Three Quality of Recovery Scales. Anesthesiology. 2016 Jul;125(1):39-45. doi: 10.1097/ALN.0000000000001158. PMID 27159009